CLINICAL TRIAL: NCT05891574
Title: Influence and Relationships Between Square-stepping Exercise and Brain Activation, Cognitive Function, Physical Performance in Healthy Older Adults
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Ray-Yau Wang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: NYCU112078AE
Record Dates: First submitted 2023-05-15; First posted 2023-06-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2023-06

CONDITIONS: Older Adults; Age Problem
Keywords: older adults; square-stepping exercise; brain activation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- healthy older adults: * Age between 65 and 90 years
  * No frailty indicated by Fried frailty criteria
  * Mini-mental state examination score equals to or more than 24, and Montreal Cognitive Assessment score equals to or more than 26
  * Ability to walk independently for 1 min

SUMMARY:
Background and purposes: Square-stepping exercise (SSE) has been proved to be an effective intervention for motor and cognitive function in older adults. However, the underlying mechanism of SSE still remains undetermined. Therefore, the aim of this study is to elucidate the possible mechanism of SSE in healthy older adults.

Methods: This is a cross-sectional study. Inclusion criteria are: (1) age between 65 and 90 years, (2) no frailty indicated by Fried frailty criteria, (3) mini-mental state examination score≧24 and Montreal Cognitive Assessment score≧26, (4) ability to walk independently for 1 min. Brain activation differences between SSE patterns and usual walking, as well as relationships between brain activity, cognitive function, physical performance and SSE performance will be examined. This study will address both cognitive and motor aspects of possible mechanism in SSE. SPSS version 25.0 (SPSS Inc., Chicago, IL, USA) will be used to analyze the collected data in this study. One-way ANOVA with repeated measures is used to evaluate the differences in brain activation among usual walking, SSE-pattern 1, and SSE-pattern 2, with Bonferroni test for post hoc analysis. The Pearson correlation coefficient will be used to establish the relationships between brain activity and SSEs performance, between cognitive function and SSEs performance, and between motor function and SSEs performance. The significant level is set at p< .05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 90 years
* No frailty indicated by Fried frailty criteria
* Mini-mental state examination score equals to or more than 24, and Montreal Cognitive Assessment score equals to or more than 26
* Ability to walk independently for 1 min

Exclusion Criteria:

* Central nervous system disorders (such as stroke, Parkinson's disease, spinal cord injury)
* Any unstable physical condition, psychiatric disorder, and other neurological disorder, or diagnosed with learning disability which may affect participating this study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy older adults
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Brain activity | at the enrollment (1 day)
  The brain (bilateral PFC, PMC, SMA) activity indicated by brain oxygenation will be measured by a wearable functional near-infrared spectroscopy system under 3 conditions: usual walking, SSE-pattern 1 (SSE1), and SSE-pattern 2 (SSE2).
  * Usual walking: participants walk back and forth at their comfortable speed on a 25-m walkway for 1 min.
  * SSE1: participants perform SSE pattern 1 on the SSE mat at their comfortable speed, and repeat the pattern for 1 min.
  * SSE2: participants perform SSE pattern 2 on the SSE mat at their comfortable speed, and repeat the pattern for 1 min.

SECONDARY OUTCOMES:
SSE performance | at the enrollment (1 day)
  The number of the correct steps that participants complete in 1 min during SSEs will be recorded. The average of the two trials for each pattern will be calculated as SSE performance for data analysis
Montreal Cognitive Assessment | at the enrollment (1 day)
  The MoCA Taiwanese Version is used to evaluate global cognitive function. It consists of eight cognitive domains, including visuospatial/ executive function, naming, memory, attention, language, abstraction, delayed recall, orientation.
Trail Making Test | at the enrollment (1 day)
  The Trail Making Test (TMT) consists part A and B, and is one of the most widely used test for executive function especially in attention, sequencing and shifting domains.
Stroop Color and Word Test | at the enrollment (1 day)
  The Stroop Color and Word Test (SCWT) is used to measure executive function especially the selective attention with high test-retest reliability of 0.91. During the test, subject is asked to (1) name the word in congruent color and (2) name the color of the ink in which incongruent color words are printed. The numbers of correct answers within 45 seconds are recorded, with the congruent and incongruent part scored separately.
Digit span test | at the enrollment (1 day)
  A subtest in Wechsler Adult Intelligence Scale Revised and is commonly used for testing attention and working memory with the test-retest reliability of 0.83. The test is composed of forward span and backward span. In forward recall, participants have to repeat the exact sequence that assessor read out. In backward span, after the forward span was completed, the participants have to repeat the sequence in reverse. The sequence ranges from 3-digit to 9-digit for forward, and 2-digit to 8-digit for backward. The total score will be the summation of forward and backward.
Timed up and go test | at the enrollment (1 day)
  The timed up and go test (TUG) is used to evaluate dynamic balance and functional mobility (ICC=0.98)62. The participant is instructed to stand up from a chair, walk as fast as possible for 3 meters, turn, walk back to the chair, and sit down. The time needed to complete the test will be recorded. The test will be repeated twice, with a 30-second rest in between, and the average will be analyzed.
Berg balance scale | at the enrollment (1 day)
  Berg-balance scale (BBS) is a 14-item measurement of balance and fall risk with test and retest reliability of 0.886. Each item is scored on a 5-point scale, ranging from 0 to 4. Total score of BBS ranges from 0 to 56.
Five times sit to stand test | at the enrollment (1 day)
  The five times sit to stand test (FSST) is used to indicate the lower extremity strength with test and retest reliability of 0.89. Participant is instructed to fold arms across chest, and performs sit-to-stand five times as quickly as possible. The test will be done twice, with a 30-second rest in between, and average time spent of the two trials will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No